CLINICAL TRIAL: NCT06392594
Title: Performance of Xpert MTB/RIF and XDR Assay for Diagnosis of Pulmonary Tuberculosis.
Brief Title: Performance of Xpert MTB/RIF and XDR Assay for Diagnosis of Pulmonary Tuberculosis and Resistant Pulmonary TB
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Esmat Mohamed Kotb, resident doctor of pulmonologist, Assiut University
Other Study IDs: Pulmonary Tuberculosis xpert
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: xpert MTB , XDR assay — To determine how accurate Xpert MTB/RIF and XDR for diagnosis of pulmonary TB and Rifampicin resistance

SUMMARY:
To determine how accurate Xpert MTB/RIF and XDR for diagnosis of pulmonary TB and Rifampicin resistance

DETAILED DESCRIPTION:
Tuberculosis (TB) is one of the major public health threats, competing with the human immunodeficiency virus (HIV) as the cause of death due to infectious diseases worldwide.

Tuberculosis (TB) is the leading cause of death by a single pathogen worldwide. In 2019, 1.2 million people died from TB among HIV-negative patients, 208 000 among HIV-positive patients and 10 million were estimated to have fallen sick, although only 70% were diagnosed The gap between TB notifications and estimated existing cases is still unacceptable. The low TB case detection rate in many high-burden settings urgently demands effective strategies and tools to identify TB patients and ensure their linkage to healthcare

MDR Multidrug-resistant tuberculosis (MDR-TB), caused by Mycobacterium tuberculosis that is resistant to both isoniazid and rifampicin with or without resistance to other drugs

* According to current World Health Organization and the International Union Against Tuberculosis and Lung Disease estimates, the median prevalence of MDR-TB has been 1.1% in newly diagnosed patients. The proportion, however, is considerably higher (median prevalence, 7%) in patients who have previously received anti-TB treatment.
* XDR tuberculosis is caused by a strain of Mycobacterium tuberculosis resistant to isoniazid and rifampin (which defines MDR tuberculosis) in addition to any fluoroquinolone and at least one of the three following injectable drugs: capreomycin, kanamycin, and amikacin

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with respiratory symptoms suggestive of pulmonary T.B 2. Patients who were able to collect a sputum sample were included in the study 3. Patients with positive xpert MTB/RIF for XDR assay

Exclusion Criteria:

* Patients who were unable to collect a sputum sample Patient with negative xpert MTB/RIF for XDR assay Patients with extrapulmonary tb Patients with positive culture for MOTT

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with respiratory symptoms suggestive of pulmonary T.B like productive cough for >3 weeks, cough of any duration accompanied by constitutional symptoms (fever for at least 3 days, night sweats or weight loss of at least 3 kg in the previous month), or hemoptysis with radiological finding suggestive of pulmonary tb
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2024-04-23 (Estimated); Primary Completion 2025-04-23 (Estimated); Study Completion 2025-05-23 (Estimated)

PRIMARY OUTCOMES:
To detect the performance of xpert MTB/RIF for detection of pulmonary tuberculosis and detection of rifampicin resistant • to detect the diagnostic accuracy of XDR in diagnosis of INH and rifampicin resistance in positive cases of xpert MTB /RIF | baseline
  All Patients with respiratory symptoms suggestive of pulmonary TB will go for • Sputum for
  * acid fast bacilli
  * culture (the gold standard )
  * Gene xpert or ultra expert
  * XDR (For positive gene xpert or ultra xpert to detect the accuracy of gene xpert in diagnosis of pulmonary tuberculosios and rifampicin resistant

SECONDARY OUTCOMES:
To assess the frequency of Xpert Ultra trace positive results . to investigate the effect of smear positive and smear negative on test accuracy | baseline
  to know the accuracy of gene xpert in related to sputum sample of acid fast bacilli